CLINICAL TRIAL: NCT02998216
Title: Pelvic Floor Symptoms and Patients´ Satisfaction After Bilateral Sacrospinous Fixation for the Primary Treatment of Pelvic Organ Prolapse ICS-POPQ Stage IV: A Prospective Observational Study
Brief Title: Pelvic Floor Symptoms After Bilateral Sacrospinous Fixation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 442/2016BO2
Record Dates: First submitted 2016-11-11; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bilateral sacrospinous fixation — Bilateral sacrospinous vaginal suspension
  Other Names: Bilateral sacrospinous vaginal suspension

SUMMARY:
This study aims to the assessment of pelvic floor symptoms and patients´ satisfaction after bilateral sacrospinous fixation for the primary treatment of pelvic organ prolapse stage IV.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* pelvic organ prolapse ICS-POPQ Stage IV, with or without uterus
* signed informed consent

Exclusion Criteria:

* gynecologic surgery in the three past months before planned surgery
* history of prolapse surgery
* participation in another study
* need to simultaneously perform other surgical procedures (i.e. rectopexy)
* ongoing chemotherapy of treatment with immunosuppressant drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female patients who are planned to receive a bilateral sacrospinous fixation as a treatment for pelvic organ prolapse Stage IV will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of pelvic floor symptoms | Twelve months
  Using the validated Germen Pelvic Floor Questionnaire (Baessler et al, Neurourol Urodynam 2004)

SECONDARY OUTCOMES:
Anatomical outcome / Prolapse stage after surgery | Twelve months
  Using the POP-Q classification tool of the International Continence Society (Bump RC et al, Am J Obstet Gynecol 1996)
Changes in quality of life | Twelve months
  Germen Pelvic Floor Questionnaire (Baessler et al, Neurourol Urodynam 2004)
Changes in sexual activity | Twelve months
  Germen Pelvic Floor Questionnaire (Baessler et al, Neurourol Urodynam 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Christl Reisenauer, Professor, Principal Investigator — Universitys Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kavvadias T, Schoenfisch B, Brucker SY, Reisenauer C. Anatomical and functional outcomes after hysterectomy and bilateral sacrospinous ligament fixation for stage IV uterovaginal prolapse: a prospective case series. BMC Urol. 2020 Aug 19;20(1):126. doi: 10.1186/s12894-020-00694-3. PMID 32814553